CLINICAL TRIAL: NCT00557440
Title: A Multi-center, Randomized, Double-blind, Double Dummy, Placebo and Active Controlled Crossover Study, to Investigate the 24 Hour FEV1 Profile of a Single Dose of QMF TWISTHALER Device in Adult Patients With Persistent Asthma
Brief Title: Investigation of the 24 Hour Forced Expiratory Flow in 1 Second (FEV1) Profile of a Single Dose of Indacaterol/Mometasone Delivered Via the TWISTHALER® Device in Adult Patients With Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQMF149A2202
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Results first posted 2013-03-21 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2009-04

CONDITIONS: Asthma
Keywords: Asthma; QMF; Indacaterol; Mometasone
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination; Mometasone Furoate; QMF149; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Ind/M - FP/Salm - Pbo (Experimental): In Treatment Period 1 (Days 1 & 2) participants received indacaterol/mometasone (Ind/M) 500/400 μg via the TWISTHALER device (2 inhalations of 250/200 μg) in the evening and placebo to fluticasone/salmeterol via multi-dose dry powder inhaler (MDDPI), one inhalation in the evening and one inhalation the following morning.
  In Treatment Period 2 (Days 8 & 9) participants received 2 inhalations of placebo to indacaterol/mometasone via the TWISTHALER device in the evening and fluticasone/salmeterol (FP/Salm) 250/50 μg via MDDPI, one inhalation in the evening and one inhalation the following morning.
  In Treatment Period 3 (Days 15 & 16) participants received 2 inhalations of placebo (Pbo) to indacaterol/mometasone via the TWISTHALER device in the evening and placebo to fluticasone/salmeterol via MDDPI, one inhalation in the evening and one inhalation the following morning.
  Each treatment period was separated by a 6-day washout period.
  Interventions: Drug: fluticasone propionate/salmeterol; Drug: indacaterol maleate / mometasone furoate; Drug: placebo to indacaterol/mometasone; Drug: placebo to fluticasone propionate/salmeterol
- FP/Salm - Pbo - Ind/M (Experimental): In Treatment Period 1 (Days 1 & 2) participants received 2 inhalations of placebo to indacaterol/mometasone via the TWISTHALER device in the evening and fluticasone/salmeterol (FP/Salm) 250/50 μg via MDDPI, one inhalation in the evening and one inhalation the following morning.
  In Treatment Period 2 (Days 8 & 9) participants received 2 inhalations of placebo to indacaterol/mometasone via the TWISTHALER device in the evening and placebo to fluticasone/salmeterol via MDDPI, one inhalation in the evening and one inhalation the following morning.
  In Treatment Period 3 (Days 15 & 16) participants received indacaterol/mometasone (Ind/M) 500/400 μg via the TWISTHALER device (2 inhalations of 250/200 μg) in the evening and placebo to fluticasone/salmeterol via MDDPI, one inhalation in the evening and one inhalation the following morning.
  Each treatment period was separated by a 6-day washout period.
  Interventions: Drug: fluticasone propionate/salmeterol; Drug: indacaterol maleate / mometasone furoate; Drug: placebo to indacaterol/mometasone; Drug: placebo to fluticasone propionate/salmeterol
- Pbo - Ind/M - FP/Salm (Experimental): In Treatment Period 1 (Days 1 & 2) participants received 2 inhalations of placebo (Pbo) to indacaterol/mometasone via the TWISTHALER device in the evening and placebo to fluticasone/salmeterol via MDDPI, one inhalation in the evening and one inhalation the following morning.
  In Treatment Period 2 (Days 8 & 9) participants received indacaterol/mometasone (Ind/M) 500/400 μg via the TWISTHALER device (2 inhalations of 250/200 μg) in the evening and placebo to fluticasone/salmeterol via MDDPI, one inhalation in the evening and one inhalation the following morning.
  In Treatment Period 3 (Days 15 & 16) participants received 2 inhalations of placebo to indacaterol/mometasone via the TWISTHALER device in the evening and fluticasone/salmeterol (FP/Salm) 250/50 μg via MDDPI, one inhalation in the evening and one inhalation the following morning.
  Each treatment period was separated by a 6-day washout period.
  Interventions: Drug: fluticasone propionate/salmeterol; Drug: indacaterol maleate / mometasone furoate; Drug: placebo to indacaterol/mometasone; Drug: placebo to fluticasone propionate/salmeterol

INTERVENTIONS:
Drug: fluticasone propionate/salmeterol — Fluticasone propionate/salmeterol 250/50 μg twice daily delivered via MDDPI.
  Other Names: Advair®; Seretide®
Drug: indacaterol maleate / mometasone furoate — Indacaterol maleate / mometasone furoate 500/400 μg once daily delivered via the TWISTHALER device.
  Other Names: QMF149
Drug: placebo to indacaterol/mometasone — Placebo to indacaterol maleate/mometasone furoate delivered via the TWISTHALER device.
Drug: placebo to fluticasone propionate/salmeterol — Placebo to fluticasone propionate / salmeterol delivered via MDDPI.

SUMMARY:
This study is designed to provide data about the 24 hours FEV1 profile, safety and tolerability of indacaterol/mometasone TWISTHALER device compared to placebo and using fluticasone/salmeterol as an active control.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult patients aged 18-75 years (inclusive), who have signed an Informed Consent Form prior to initiation of any study-related procedure,
* Patients with persistent asthma, diagnosed according to Global Initiative for Asthma (GINA) guidelines (National Institute of Health, National Heart, Lung and Blood Institute, 2006) and who additionally meet the following criteria:

  * Patients receiving daily treatment with inhaled corticosteroid up to the maximum dose per day indicated in the product label, in a stable regimen for the month prior to Visit 1.
  * Patients with an FEV1 at Visit 1 ≥50% of predicted normal.
  * Patients who demonstrate an increase of ≥ 12% and ≥ 200 mL in FEV1 over their pre-bronchodilator.

Exclusion Criteria:

* Pregnant women, nursing mothers, or females of childbearing potential, regardless of whether or not sexually active, if they are not using a reliable form of contraception.
* Patients who have used tobacco products within the 6 months period prior to Visit 1, or who have a smoking history of greater than 10 pack years.
* Patients diagnosed with Chronic Obstructive Pulmonary disease (COPD) as defined by the GOLD guidelines (Global Initiative for Chronic Obstructive Lung Disease 2006).
* Patients with seasonal allergy whose asthma is likely to deteriorate during the study period.
* Patients who have had an acute asthma attack/exacerbation requiring hospitalization in the 6 months prior to Visit 1.
* Patients who have had an acute asthma attack / exacerbation requiring an emergency room visit within 6 weeks prior to Visit 1 or at any time between Visit 1 and Visit 2.
* Patients who have had a respiratory tract infection within 4 weeks prior to Visit 1 or at any time between Visit 1 and Visit 2.
* Patients with a history of long QT interval syndrome or whose QT interval corrected for heart rate (QTc) interval (Bazett's) measured at Visit 1 or Visit 2 is prolonged: > 450 ms (males) or > 470 ms (females).
* Other clinically significant conditions which may interfere with the study conduct or patient safety as specified in the protocol.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma, Study Chair — Novartis Pharmaceuticals
Locations (6):
- Belgium (2):
  - Novartis Investigator Site, Aalst
  - Novartis Investigator site, Ghent
- Germany (4):
  - Novartis Investigator Site, Berlin
  - Novartis Investigator Site, Hanover
  - Novartis Investigator Site, Landsberg
  - Novartis Investigator Site, Rostock

RESULTS

PARTICIPANT FLOW:
Groups:
- Ind/M - FP/Salm - Pbo: In Treatment Period 1 (Days 1 & 2) participants received indacaterol/mometasone (Ind/M) 500/400 μg via the TWISTHALER device (2 inhalations of 250/200 μg) in the evening and placebo to fluticasone/salmeterol via multi-dose dry powder inhaler (MDDPI), one inhalation in the evening and one inhalation the following morning.
  In Treatment Period 2 (Days 8 & 9) participants received 2 inhalations of placebo to indacaterol/mometasone via the TWISTHALER device in the evening and fluticasone /salmeterol (FP/Salm) 250/50 μg via MDDPI, one inhalation in the evening and one inhalation the following morning.
  In Treatment Period 3 (Days 15 & 16) participants received 2 inhalations of placebo (Pbo) to indacaterol/mometasone via the TWISTHALER device in the evening and placebo to fluticasone/salmeterol via MDDPI, one inhalation in the evening and one inhalation the following morning.
  Each treatment period was separated by a 6-day washout period.
Period: Treatment Period 1
Arm/Group | Ind/M - FP/Salm - Pbo | FP/Salm - Pbo - Ind/M | Pbo - Ind/M - FP/Salm
Started | 12 | 12 | 13
Completed | 12 | 12 | 12
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1
Period: Treatment Period 2
Arm/Group | Ind/M - FP/Salm - Pbo | FP/Salm - Pbo - Ind/M | Pbo - Ind/M - FP/Salm
Started | 12 | 12 | 12
Completed | 12 | 12 | 12
Not Completed | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Ind/M - FP/Salm - Pbo | FP/Salm - Pbo - Ind/M | Pbo - Ind/M - FP/Salm
Started | 12 | 12 | 12
Completed | 12 | 12 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ind/M - FP/Salm - Pbo | FP/Salm - Pbo - Ind/M | Pbo - Ind/M - FP/Salm | Total
Number analyzed (Participants) | 12 | 12 | 13 | 37
Age Continuous [Mean (Standard Deviation); unit: years] | 40.2 (15.37) | 50.5 (12.00) | 52.5 (10.46) | 47.9 (13.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 7 | 15
  Male | 7 | 9 | 6 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Period Baseline to 24 Hour Post-dose (Trough) Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Change from the period baseline to 24 hour post dose trough FEV1 after 1 day of treatment was analyzed using Analysis of Covariance (ANCOVA) adjusting for treatment, period, sequence and center with period baseline as a covariate and patient nested within sequence as a random effect.
Time Frame: Pre-dose for each Treatment Period (Days 1, 8 and 15) and 24-hours post-dose for each Treatment Period (Days 2, 9 and 16).
Population: The Intent-To-Treat (ITT) population included all randomized patients who had at least one period containing a Baseline FEV1 measurement and at least one post-baseline measurement of FEV1 for the same treatment period. Patients who took rescue medication within 6 hours prior to the trough measurements were excluded from the analysis.
Measure: Least Squares Mean (Standard Error); unit: liters
Groups:
- Indacaterol/Mometasone: Participants received a single dose of indacaterol/mometasone 500/400 μg delivered via the TWISTHALER device (2 inhalations of 250/200 μg) in the evening.
- Fluticasone/Salmeterol: Participants received fluticasone/salmeterol 250/50 μg via multi-dose dry powder inhaler (MDDPI), one inhalation in the evening and one inhalation the following morning.
- Placebo: Participants received placebo to indacaterol/mometasone via the TWISTHALER device and placebo to fluticasone/salmeterol via MDDPI.
Arm/Group | Indacaterol/Mometasone | Fluticasone/Salmeterol | Placebo
Number analyzed (Participants) | 36 | 36 | 35
liters | 0.081 (0.0473) | 0.049 (0.0472) | -0.083 (0.0475)
Statistical Analysis 1: Comparison: Indacaterol/Mometasone vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA — Statistical significance (two-sided) at 5% level. p-values were not corrected for multiplicity; Treatment, period, sequence and center as fixed effects, period baseline FEV1 as a covariate, and patient nested within sequence as a random effect; LS Mean Difference = 0.165, 95% CI 2-sided [0.066 to 0.263], Standard Error of Mean 0.0492

2. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) at Single Time Points
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. FEV1 was analyzed using Analysis of Covariance (ANCOVA) adjusting for treatment, period, sequence and center with period baseline as a covariate and patient nested within sequence as a random effect.
Time Frame: 5, 30 minutes, 1, 2, 3, 4 hours, 11 hours 10 minutes, 11 hours 45 minutes, 12 hours 30 minutes, 14, 16, 18, 20, 22 hours, 23 hours 10 minutes, and 23 hours 45 minutes post-dosing.
Population: Intent-to-treat population, where data were available. Patients who took rescue medication within 6 hours prior to spirometry measurements were excluded from the analysis. N indicates the number of participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Indacaterol/Mometasone | Fluticasone/Salmeterol | Placebo
Number analyzed (Participants) | 36 | 36 | 37
liters
  5 minutes [N=36, 36, 37] | 2.713 (0.0302) | 2.632 (0.0302) | 2.554 (0.0300)
  30 minutes [N=36, 36, 36] | 2.754 (0.0316) | 2.719 (0.0316) | 2.527 (0.0316)
  1 hour [N=36, 36, 36] | 2.760 (0.0350) | 2.771 (0.0350) | 2.525 (0.0350)
  2 hours [N=36, 36, 36] | 2.754 (0.0400) | 2.734 (0.0399) | 2.483 (0.0400)
  3 hours [N=36, 36, 36] | 2.728 (0.0411) | 2.724 (0.0410) | 2.425 (0.0411)
  4 hours [N=36, 36, 35] | 2.705 (0.0434) | 2.669 (0.0434) | 2.376 (0.0437)
  11 hours 10 minutes [N=36, 35, 34] | 2.685 (0.0496) | 2.570 (0.0499) | 2.295 (0.0505)
  11 hours 45 minutes [N=36, 35, 32] | 2.628 (0.0492) | 2.518 (0.0495) | 2.276 (0.0509)
  12 hours 30 minutes [N=36, 35, 32] | 2.667 (0.0437) | 2.659 (0.0440) | 2.359 (0.0453)
  14 hours [N=36, 35, 32] | 2.766 (0.0433) | 2.779 (0.0436) | 2.485 (0.0448)
  16 hours [N=36, 35, 31] | 2.720 (0.0493) | 2.681 (0.0497) | 2.454 (0.0515)
  18 hours [N=35, 36, 33] | 2.729 (0.0395) | 2.717 (0.0389) | 2.513 (0.0398)
  20 hours [N=35, 36, 34] | 2.725 (0.0475) | 2.707 (0.0467) | 2.479 (0.0475)
  22 hours [N=35, 36, 34] | 2.674 (0.0493) | 2.695 (0.0485) | 2.487 (0.0493)
  23 hours 10 minutes [N=35, 36, 35] | 2.696 (0.0517) | 2.676 (0.0510) | 2.530 (0.0513)
  23 hours 45 minutes [N=36, 36, 34] | 2.686 (0.0459) | 2.640 (0.0458) | 2.523 (0.0464)
  24 hours post-dose trough [N=36, 36, 35] | 2.689 (0.0473) | 2.656 (0.0472) | 2.524 (0.0475)

3. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Standardized Area Under the Curve (AUC) Between Baseline (Pre-dose) and 24 Hours Post-dose
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. FEV1 was measured pre-dose and up to 24 hours post-dose. The FEV1 standardized area under the curve (AUC) was analyzed for four time intervals:
  * Baseline (pre-dose) to 4 hours (hr) post-dosing;
  * Baseline (pre-dose) to 23 hours, 45 minutes (min) post-dosing;
  * 11 hours, 10 minutes to 12 hours, 30 minutes post-dosing;
  * 11 hours, 10 minutes to 23 hours, 45 minutes post-dosing.
  AUC for FEV1 was analyzed using Analysis of Covariance adjusting for treatment, period, sequence and center with period baseline as a covariate and patient nested within sequence as a random effect.
Time Frame: Pre-dose, 5, 30 minutes, 1, 2, 3, 4 hours, 11 hours 10 minutes, 11 hours 45 minutes, 12 hours 30 minutes, 14, 16, 18, 20, 22 hours, 23 hours 10 minutes, and 23 hours 45 minutes post-dosing.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Indacaterol/Mometasone | Fluticasone/Salmeterol | Placebo
Number analyzed (Participants) | 36 | 36 | 37
liters
  Baseline to 4 hours [N=36, 36, 37] | 2.730 (0.0327) | 2.713 (0.0327) | 2.469 (0.0326)
  Baseline to 23 hours, 45 minutes [N=36, 36, 37] | 2.718 (0.0376) | 2.679 (0.0376) | 2.430 (0.0374)
  11 hr, 10 min to 12 hr, 30 min [N=36, 35, 34] | 2.667 (0.0443) | 2.585 (0.0445) | 2.314 (0.0451)
  11 hr, 10 min to 23 hr, 45min [N=36, 36, 36] | 2.726 (0.0435) | 2.696 (0.0435) | 2.470 (0.0436)

4. Secondary Outcome: Time to Peak Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Time to peak FEV1 is calculated in minutes from the time of inhalation of study drug to the time of the peak FEV1 during the first 4 hours post-dose.
  Time to peak FEV1 is based on log-transformed analysis of variance adjusted for treatment, period, sequence and center, with patient nested within sequence as a random effect. Geometric Mean was obtained by taking anti-logs of the adjusted means from the model and standard error was calculated using the delta method.
Time Frame: Up to 4 hours post-dose
Population: Intent-to-treat population, where data were available. Patients who took rescue medication within 6 hours prior to spirometry measurements were excluded from the analysis.
Measure: Geometric Mean (Standard Error); unit: minutes
Arm/Group | Indacaterol/Mometasone | Fluticasone/Salmeterol | Placebo
Number analyzed (Participants) | 36 | 36 | 37
minutes | 87.4 (16.98) | 67.7 (13.16) | 22.3 (4.30)

5. Secondary Outcome: Forced Vital Capacity (FVC) at Single Time Points
Description: Vital capacity is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible.
  FVC was analyzed using ANCOVA adjusting for treatment, period, sequence and center with period baseline as a covariate and patient nested within sequence as a random effect.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Indacaterol/Mometasone | Fluticasone/Salmeterol | Placebo
Number analyzed (Participants) | 36 | 36 | 37
liters
  5 minutes [N= 36, 36, 37] | 3.917 (0.0333) | 3.880 (0.0333) | 3.830 (0.0331)
  30 minutes [N= 36, 36, 36] | 3.946 (0.0338) | 3.933 (0.0338) | 3.839 (0.0338)
  1 hour [N= 36, 36, 36] | 3.945 (0.0337) | 3.955 (0.0337) | 3.808 (0.0337)
  2 hours [N= 36, 36, 36] | 4.080 (0.1074) | 3.899 (0.1073) | 3.742 (0.1073)
  3 hours [N= 36, 36, 36] | 3.925 (0.0390) | 3.923 (0.0390) | 3.708 (0.0391)
  4 hours [N= 36, 36, 35] | 3.857 (0.0438) | 3.861 (0.0438) | 3.665 (0.0442)
  11 hours 10 minutes [N= 36, 35, 34] | 3.896 (0.0569) | 3.828 (0.0573) | 3.632 (0.0581)
  11 hours 45 minutes [N= 36, 35, 32] | 3.837 (0.0549) | 3.736 (0.0553) | 3.607 (0.0570)
  12 hours 30 minutes [N= 36, 35, 32] | 3.833 (0.0496) | 3.841 (0.0500) | 3.680 (0.0518)
  14 hours [N= 36, 35, 32] | 3.918 (0.0506) | 3.894 (0.0510) | 3.759 (0.0528)
  16 hours [N= 36, 35, 31] | 3.896 (0.0524) | 3.787 (0.0528) | 3.737 (0.0551)
  18 hours [N= 35, 36, 33] | 3.893 (0.0462) | 3.866 (0.0455) | 3.784 (0.0466)
  20 hours [N= 35, 36, 34] | 3.903 (0.0499) | 3.848 (0.0492) | 3.764 (0.0499)
  22 hours [N= 35, 36, 34] | 3.865 (0.0453) | 3.906 (0.0446) | 3.764 (0.0453)
  23 hours 10 minutes [N= 35, 36, 35] | 3.870 (0.0519) | 3.866 (0.0512) | 3.808 (0.0516)
  23 hours 45 minutes [N=36, 36, 34] | 3.866 (0.0509) | 3.825 (0.0509) | 3.817 (0.0516)

ADVERSE EVENTS:
Arm/Group | Indacaterol/Mometasone | Fluticasone/Salmeterol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/37
Other Adverse Events (participants affected / at risk) | 2/36 | 1/36 | 2/37
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol/Mometasone (N=36) | Fluticasone/Salmeterol (N=36) | Placebo (N=37)
Headache (Nervous system disorders) | 2 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.